CLINICAL TRIAL: NCT06502301
Title: Evaluation of Balance With Computerized Posturography Device and Clinical Tests in Patients With Postmenopausal Osteoporosis
Brief Title: How Vertebral Fractures Effect Balance In Postmenopausal Women
Status: Completed | Type: Observational
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Dilara Okutan Kuzu, Principal Investigator, Istanbul University - Cerrahpasa
Other Study IDs: 89403766-604.01.02-136365
Record Dates: First submitted 2024-07-09; First posted 2024-07-16 (Actual); Last update posted 2024-07-16 (Actual); Status verified 2024-07

CONDITIONS: Postmenopausal Osteoporosis; Vertebral Fracture; Fracture of Vertebra; Fall
Keywords: balance; computed static posturography; fall; FRAX; vertebral fracture
MeSH Terms: conditions — Osteoporosis, Postmenopausal; Spinal Fractures | interventions — Cross-Sectional Studies

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Postmenopausal women with vertebral fractures: Thoracolumbar radiograph, computed static posturography, fracture risk assessment tool (FRAX) scores, Dual-energy x-ray absorptiometry (DXA) measurements, serum 25(OH)D values, tandem test, timed up and go test (TUG), Berg balance scale (BBS) were performed.
  Interventions: Other: Cross-sectional study
- Postmenopausal women without vertebral fractures: Thoracolumbar radiograph, computed static posturography, fracture risk assessment tool (FRAX) scores, Dual-energy x-ray absorptiometry (DXA) measurements, serum 25(OH)D values, tandem test, timed up and go test (TUG), Berg balance scale (BBS) were performed.
  Interventions: Other: Cross-sectional study

INTERVENTIONS:
Other: Cross-sectional study — This is not intervention study.

SUMMARY:
Osteoporosis is defined as low bone mineral density caused by altered bone microstructure, ultimately predisposing patients to fragility fractures. Osteoporotic fractures lead to a significant decrease in quality of life, increasing morbidity, mortality, and disability. Vertebral fracture may cause sagittal imbalance which leading to postural instability and becomes a possible risk factor for falls. The cause of balance problems in osteoporotic patients is multifactorial including increased thoracic kyphosis and postural sway, however the exact relationship between vertebral fractures and balance remains unclear. The aim of the study is; to evaluate the effect of the presence of a vertebral fracture on balance and physical performance and its contribution to fall and fracture risk in patients with postmenopausal osteoporosis.

DETAILED DESCRIPTION:
Osteoporosis is a metabolic bone disease characterized by low bone mass, deterioration of bone tissue, and disruption of bone microarchitecture . It is known that the incidence of vertebral fractures in women with osteoporosis increases especially after the age of 50. In the United States, one in four women older than 50 years suffers at least one osteoporosis-related vertebral compression fractures. Approximately one-third of vertebral fractures become symptomatic . Vertebral fracture may cause increased dorsal kyphosis and, the center of gravity of the body moves forward. Impaired postural stability is associated with fall risk and functional disability .

Many authors argue that the osteoporotic vertebral fractures are associated with an increase in the thoracic curve. There are studies revealing that hyperkyphosis may be a clinically useful marker for history of vertebral fracture and also a risk factor for a new vertebral fracture. Postmenopausal women with vertebral fracture have a 4-fold increased risk of new fractures compared to whom without spinal fracture. Recent vertebral fractures have a strong impact on daily living activities and are significant predictors of poor performance in functional status of the patient. However this triangle among vertebral fractures, kyphosis and balance has not been well documented in the literature.

The vertebral fracture cascade phenomena raises the possibility that multiple factors, such as spinal characteristics, vertebral alignment, spinal curvature, and spinal loads, as well as low bone mineral density, may have an impact on falls and fractures. Vertebral fracture may cause sagittal imbalance which leading to postural instability and becomes a possible risk factor for falls. Especially in osteoporotic elderly; falls are associated with high morbidity and mortality. However the effect of a vertebral fracture, as a preventable risk factor on balance impairment has not been studied sufficiently. In this study, we aimed to assess the effect of the presence of a vertebral fracture on balance and physical performance and its additional contribution to fall and fracture risk in patients with postmenopausal osteoporosis.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged 50 years or older
2. Diagnosis of postmenopausal osteoporosis according to WHO (World Health Organization) criteria and/or osteoporotic vertebral fractures

Exclusion Criteria:

1. A history of neurological and/or vestibular system disease
2. Using a medication that may affect balance and proprioception
3. The presence of a psychotic disorder
4. A history of lower extremity surgery in the last 6 months

Min Age: 50 Years | Sex: Female
Age Groups: Adult, Older Adult
Study Population: 95 patients, at the age of 50 and above with postmenopausal osteoporosis and/or osteoporotic vertebral fractures according to WHO criteria were included in this study.
Sampling Method: Non-Probability Sample
Enrollment: 95 (Actual)
Dates: Start 2020-11-01 (Actual); Primary Completion 2021-02-28 (Actual); Study Completion 2021-02-28 (Actual)

PRIMARY OUTCOMES:
Computed static posturography | Baseline
  Computerized systems play a crucial role in the quantitative and dynamic evaluation of balance function. The Tetrax device, a computerized static posturography system developed by Sunlight Medical Ltd, Israel, was utilized in our study. This device is valuable for both diagnosis and treatment purposes, offering quantitative assessment of balance. Participants underwent evaluation using the Tetrax device, which involved 32-second measurements in eight different positions. The device calculates several parameters including the Stability Index (SI), Fall Index (FI), and Fourier frequencies, providing objective measures of balance function.

SECONDARY OUTCOMES:
Timed and go test (TUG) | Baseline
  TUG is the shortest, simplest and probably the most reliable clinical balance test. There is a significant relationship between TUG times and functional mobility level. A recent systematic review showed that TUG is clinically applicable and reliable across multiple populations. In our study, patients were instructed to begin in a seated position, then stand up, walk a distance of three meters to cross a line on the ground, turn around, walk back, and sit down again. The time taken to complete this task was measured using a chronometer.
Berg balance scale (BBS) | Baseline
  Berg balance scale (BBS) was originally developed for the assessment of postural control, and is widely used in many areas of rehabilitation. There are 14 items in the scale, like commonly performing in daily activities sitting and standing balance, transfers, turning, and retrieving objects from the floor. BBS has high specificity and low sensitivity in patients at increased risk of falls. We used Turkish version of BBS whose reliability and validity in the Turkish language have been demonstrated.
Tandem stance test | 10 second
  Static balance was assessed using the tandem stance test. Patients were asked to maintain tandem stance position for 10 seconds without moving, with one foot's toe directly in front of the heel of the other foot. The test outcomes were recorded as either successful or unsuccessful. Participants unable to maintain the stance for the full 10 seconds were deemed unsuccessful, indicating an increased risk of falling.
Tandem gait test | Baseline
  Dynamic balance was evaluated using the tandem gait test. The patients were asked to take 10 consecutive steps with the toe of one toe and the heel of the other foot aligned. Patients who completed 10 serial steps were considered successful, while inability to complete the steps indicated an unsuccessful test.
Fracture Risk Assessment tool (FRAX) | Baseline
  The fracture risk assessed with the FRAX tool (Fracture Risk Assessment tool). The clinical fracture risk factors of the patients were also questioned. The 10-year major osteoporotic and hip fracture risks of the patients were calculated by using the BMD (g/cm2) of the femoral neck.
Dual-energy x-ray absorptiometry measurements | Baseline
  Bone density measurements were performed using the same DXA device for all participants (n =95) (Hologic QDR 4500SL (S/N 45624) (Bedford, MA). Osteoporosis was defined as a T-score of -2.5 SD or lower in any patient. The areal BMD (aBMD) (g/cm2) and T-score of the femoral neck (FN) and lumbar spine (LS) were used in the analyses.

CONTACTS AND LOCATIONS:
Overall Officials: Sansin Tuzun, Study Director — Istanbul University - Cerrahpasa; Dilara Okutan Kuzu, Principal Investigator — Istanbul University - Cerrahpasa; Rana Kaynar Terlemez, Study Chair — Istanbul University - Cerrahpasa; Deniz Palamar Kadioglu, Study Chair — Istanbul University - Cerrahpasa
Locations (1):
- Istanbul University-Cerrahpasa, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cosman F, de Beur SJ, LeBoff MS, Lewiecki EM, Tanner B, Randall S, Lindsay R; National Osteoporosis Foundation. Clinician's Guide to Prevention and Treatment of Osteoporosis. Osteoporos Int. 2014 Oct;25(10):2359-81. doi: 10.1007/s00198-014-2794-2. Epub 2014 Aug 15. PMID 25182228
- [Background] Sozen T, Ozisik L, Basaran NC. An overview and management of osteoporosis. Eur J Rheumatol. 2017 Mar;4(1):46-56. doi: 10.5152/eurjrheum.2016.048. Epub 2016 Dec 30. PMID 28293453
- [Background] Wang LY, Liaw MY, Huang YC, Lau YC, Leong CP, Pong YP, Chen CL. Static and dynamic balance performance in patients with osteoporotic vertebral compression fracture. J Back Musculoskelet Rehabil. 2013;26(2):199-205. doi: 10.3233/BMR-130369. PMID 23640322
- [Background] Lems WF. Clinical relevance of vertebral fractures. Ann Rheum Dis. 2007 Jan;66(1):2-4. doi: 10.1136/ard.2006.058313. PMID 17178757
- [Background] Lynn SG, Sinaki M, Westerlind KC. Balance characteristics of persons with osteoporosis. Arch Phys Med Rehabil. 1997 Mar;78(3):273-7. doi: 10.1016/s0003-9993(97)90033-2. PMID 9084349
- [Background] Katzman WB, Vittinghoff E, Kado DM, Lane NE, Ensrud KE, Shipp K. Thoracic kyphosis and rate of incident vertebral fractures: the Fracture Intervention Trial. Osteoporos Int. 2016 Mar;27(3):899-903. doi: 10.1007/s00198-015-3478-2. Epub 2016 Jan 18. PMID 26782685
- [Background] Huang MH, Barrett-Connor E, Greendale GA, Kado DM. Hyperkyphotic posture and risk of future osteoporotic fractures: the Rancho Bernardo study. J Bone Miner Res. 2006 Mar;21(3):419-23. doi: 10.1359/JBMR.051201. Epub 2005 Dec 5. PMID 16491290
- [Background] Huang C, Ross PD, Wasnich RD. Vertebral fracture and other predictors of physical impairment and health care utilization. Arch Intern Med. 1996 Nov 25;156(21):2469-75. PMID 8944740
- [Background] Briggs AM, Greig AM, Wark JD. The vertebral fracture cascade in osteoporosis: a review of aetiopathogenesis. Osteoporos Int. 2007 May;18(5):575-84. doi: 10.1007/s00198-006-0304-x. Epub 2007 Jan 6. PMID 17206492